CLINICAL TRIAL: NCT00867659
Title: The Role of Cetrotide Acetate in Prevention of Ovarian Hyperstimulation Syndrome in Oocyte Donors
Brief Title: The Role of Cetrotide Acetate in Prevention of Ovarian Hyperstimulation Syndrome (OHSS) in Oocyte Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Fady I. Sharara, M.D, Medical Director, Virginia Center for Reproductive Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VCRM2
Record Dates: First submitted 2009-03-21; First posted 2009-03-24 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: ovarian hyperstimulation syndrome; cetrotide acetate; GnRH antagonist; oocyte donors
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetrotide acetate (Experimental): oocyte donors will receive cetrotide acetate on the day of oocyte retrieval. The incidence of OHSS will be assessed.
  Interventions: Drug: Cetrotide acetate

INTERVENTIONS:
Drug: Cetrotide acetate — cetrotide acetate is a GnRH antagonist. The dose is 3 mg once on the day of oocyte retrieval.

SUMMARY:
This pilot study aims to address whether the prophylactic use of Cetrorelix Acetate after a long gonadotropin-releasing hormone (GnRH) agonist protocol post-hCG (human chorionic gonadotropin) administration can significantly reduce the incidence of OHSS in oocyte donors.

DETAILED DESCRIPTION:
With varying complications, OHSS is an iatrogenic condition cause by ovarian stimulation. Classified as mild, moderate, or severe, mild OHSS is relatively common as it occurs in up to 1/3 of women undergoing ovarian stimulation. Symptoms include abdominal ascites, nausea, vomiting, increased abdominal girth and weight gain, with increasing ranges for mild to moderate. Severe OHSS occurs in 1% and includes hemodynamic instability, thrombosis, pulmonary difficulties, oliguria, and rarely death. Therefore, strategies to prevent or severely decrease the incidence of OHSS are sorely needed.

More aggressive ovarian stimulation increases the risk of OHSS, but it is not easy to predict who or who will not develop OHSS. Certain patient types, however, are considered to be at a higher risk than others, including oocyte donors. OHSS in oocyte donors manifests early, i.e. within days of oocyte retrieval, yet does not have the continued complication of pregnancy as observed in IVF patients. Therefore, as a in this vulnerable patient population, oocyte donors are ideal to study.

GnRH antagonists been most recently used in high risk patients undergoing IVF. Aside the reduction of OHSS observed after the traditional utilization of the antagonist protocol, alternative uses have also suggested favorable outcomes. Two retrospective, cohort matched studies evaluated a Ganirelix Acetate substitution in women who were at high risk for developing OHSS (E2 > 2,000 pg/ml on cycle day 6 or a projected peak E2 > 5,000 pg/ml with > 25 follicles on the day of HCG administration) after being down-regulated using GnRHa (or using a microdose flare protocol) and undergoing ovarian stimulation The GnRHa was stopped and only a low dose of hMG was continued when Ganirelix Acetate was started. The Ganirelix Acetate use resulted in an average drop of 41-49.5% in peak E2 levels. While those two studies were provocative, they were retrospective and not controlled. In the only prospective study evaluating the use of Ganirelix Acetate in the prevention of OHSS compared to coasting, the "historic" gold standard, Ganirelix Acetate resulted in a 36% drop in E2 level after one injection and a 59% drop in peak E2 after 3 days of use (46.8% required only one injection, 38.3% required two, and only 14.9% required 3 injections) as opposed to a 9% increase in E2 level 24 hours after coasting. The use of Ganirelix acetate resulted in significant decrease in OHSS risk (2.1-2.3% in the two retrospective studies, and 0% in the only prospective study vs 9-38% in prior publications) without affecting the pregnancy outcome. The mean number of Ganirelix Acetate injections was 1.74 + 0.91. Although, Ganirelix Acetate appears to be successful in lowering the OHSS risk previous to hCG administration as suggested by these studies, this pilot study questions the effect after the ovulation induction is administered. To date, no such study has asked this question.

All donors will be evaluated daily with hormonal levels (FSH, LH, E2, P, CBC, and comprehensive metabolic profile (which includes liver function tests) for at least 3 days after the oocyte retrieval. Daily weights and abdominal circumference will also be measured. All oocyte donors will also present for one last visit one week after oocyte retrieval. The incidence of OHSS will be the main outcome measured.

ELIGIBILITY:
Inclusion Criteria:

* Prospective donors with BMIs between 19 and 28,
* Those with normal FSH levels and good antral follicle counts between 19-28 years of age, AND
* Donors would have passed all the required testing as mandated by VCRM and the FDA.

Exclusion Criteria:

* Oocyte donors exceeding a BMI of > 28,
* Those with any communicable diseases,
* Those with low antral follicle counts and small ovarian volumes,
* Those with elevated FSH levels,
* Those with positive sickle cell screen or cystic fibrosis screening,
* Smokers, OR
* Donors who are unable or unwilling to follow the research protocols.

Ages: 19 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fady I Sharara, M.D, Principal Investigator — Virginia Center for Reproductive Medicine
Locations (1):
- Virginia Center for Reproductive Medicine, Reston, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fertility practice. 20 oocyte donors completed the study bettwen 2009 and 2011
Pre-assignment Details: Long acting Cetrotide acetate was used in an attempt to prevent ovarian hyperstimulation syndrome.
Groups:
- Cetrotide Acetate: oocyte donors will receive 3 mg cetrotide acetate by a single injection on the day of oocyte retrieval. The incidence of OHSS will be assessed.
Period: Overall Study
Arm/Group | Cetrotide Acetate
Started | 20 (October 2009)
Completed | 20 (January 2010)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetrotide Acetate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
incidence of ovarian hyperstimulation [Number; unit: particpants] — Incidence of OHSS will be assessed in 20 oocyte donors
  particpants | 20

OUTCOME MEASURES:

1. Primary Outcome: Volume of Ascites in the Abdomen is Indicative of the Severity of OHSS
Description: evaluate by ultrasound examination, physical examination and blood work the incidence of ovarian hyperstimulation syndrome in oocyte donors receiving a single injection of 3 mg Cetrotide Acetate.
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: cc (volume of ascites)
Groups:
- Cetrotide Acetate: oocyte donors will receive a single injection of 3 mg cetrotide acetate on the day of oocyte retrieval. The incidence of OHSS will be assessed.
Arm/Group | Cetrotide Acetate
Number analyzed (Participants) | 20
cc (volume of ascites) | 10 [0 to 90]

2. Primary Outcome: Ovarian Volumes as a Predictor of OHSS Severity
Description: ultrasound measurements of both ovaries
Time Frame: 30 days
Measure: Mean (Full Range); unit: cc
Arm/Group | Cetrotide Acetate
Number analyzed (Participants) | 20
cc | 25 [10 to 55]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cetrotide Acetate
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Only 20 donors were recruited because this was a pilot study to assess the benefit of Cetrotide acetate in oocyte donors in the prevention of ovarian hyperstimulation syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No